CLINICAL TRIAL: NCT02699866
Title: A Multi-Center, Prospective, Single Cohort, Post-Market Clinical Follow-Up (PMCF) Study to Assess Implant Survival After Insertion of Straumann® Bone Level Tapered (BLT) Implant Ø 2.9 mm in the Clinical Practice Setting
Brief Title: Implant Survival After Insertion of Bone Level Tapered (BLT) Implant Ø 2.9 mm in the Clinical Practice Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Straumann AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CR02/15
Record Dates: First submitted 2016-03-01; First posted 2016-03-04 (Estimated); Results first posted 2020-09-17 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Tooth Loss
Keywords: Small diameter implant
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BLT Implant Ø 2.9 mm (Experimental): The Straumann BLT Implants Ø 2.9 mm are available with a length of 10, 12 and 14 mm.
  Interventions: Device: BLT Implant Ø 2.9 mm

INTERVENTIONS:
Device: BLT Implant Ø 2.9 mm — Placement of Straumann BLT implants Ø 2.9 mm in central and lateral incisors in the mandible and lateral incisors in the maxilla for single tooth replacement followed by prosthetic loading.
  Other Names: Short Diameter Implant (SDI)

SUMMARY:
The Straumann Bone Level Tapered (BLT) implant Ø 2.9 mm implant was developed to allow treatment of patients with single tooth gaps of small dimensions in the lateral and central incisor positions in the mandible and in the lateral incisor positions in the maxilla. These positions are reduced-load-bearing compared to more posterior positions.

During this study performance and safety of the Straumann BLT implants Ø 2.9 mm in the clinical practice setting will be investigated.

DETAILED DESCRIPTION:
This is a multi-center, prospective, single cohort, post-market clinical follow-up (PMCF) study. The total study duration for each patient should be 12 ± 1 months.

Straumann BLT implants Ø 2.9 mm will be placed in central and lateral incisors in the mandible and lateral incisors in the maxilla for single tooth replacement, followed by provisional prosthetic loading after 6 ± 2 weeks and by final prosthetic loading 4 ± 1 months after implant placements.

In total 7 visits per patient are scheduled in this study. Implant survival, PES, implant success, bone level changes and adverse events (AEs) will be assessed.

The investigational device is a CE-(Conformité Européenne, meaning European Conformity) marked product. Straumann BLT implants Ø 2.9 mm Roxolid SLActive (sand blasted, large grit, acid etched surface) are available in lengths of 10, 12 and 14 mm.

Four centers in Germany will participate. The study and any amendments will be performed as far as possible according to International Organization for Standardization (ISO) 14155 and conform to the Declaration of Helsinki (last revision Fortaleza 2013) and local legal and regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have voluntarily signed the Informed Consent Form before any study related procedures are performed, are willing and able to attend scheduled follow-up visits and agree that the pseudonymized data are collected and analyzed.
* Patients must be males or females who are a minimum of 18 years of age.
* Patients with a minimum of 4 weeks history of edentulism in the study area, minimal interdental space and in need of a single tooth replacement with a dental implant central and lateral incisors in the mandible and lateral incisors in the maxilla (Federation Dentaire Internationale (FDI) positions 12, 22, 31, 32, 41 or 42).
* Presence of natural tooth or implants adjacent to the study implant position (single tooth gap).
* Patients with complete soft tissue coverage of the socket at implant placement.

Exclusion Criteria:

* Patients with inadequate bone volume and / or quality or metabolic bone disorder.
* Patients with local root remnants.
* Patients with inadequate wound healing capacity.
* Patients with not completed maxillary and mandibular growth.
* Patients with serious internal medical problems, uncontrolled bleeding disorders, psychoses, prolonged therapy-resistant functional disorders, xerostomia, weakened immune system, illnesses requiring periodic use of steroids or uncontrollable endocrine disorders.
* Patients with poor general state of health.
* Patients with drug or alcohol abuse.
* Patients with allergies or hypersensitivity to chemical ingredients of titanium-zirconium alloy.
* Patients with conditions or circumstances, in the opinion of the Investigator, which would prevent completion of study participation or interfere with analysis of study results, such as history of non-compliance or unreliability.
* A woman who is pregnant or planning to become pregnant at any point during the study duration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-02; Primary Completion 2019-06-30 (Actual); Study Completion 2019-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keyvan Sagheb, Dr., Principal Investigator — Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Klinik für Mund-Kiefer-Gesichtschirurgie, Plastische Operationen
Locations (5):
- Germany (5):
  - Kieferchirurgische Gemeinschaftspraxis Dr. Dr. Stroink & Kollegen, Düsseldorf
  - Medi+, Mainz
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Klinik für Mund-Kiefer-Gesichtschirurgie, Plastische Operationen, Mainz
  - Universitätsklinikum Münster, Klinik für Mund-, Kiefer- und Gesichtschirurgie, Münster
  - Kieferchirurgische Praxen Hentschel & Herrmann, Zwickau

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Steinemann SG. Titanium--the material of choice? Periodontol 2000. 1998 Jun;17:7-21. doi: 10.1111/j.1600-0757.1998.tb00119.x. No abstract available. PMID 10337309
- [Background] Gottlow J, Dard M, Kjellson F, Obrecht M, Sennerby L. Evaluation of a new titanium-zirconium dental implant: a biomechanical and histological comparative study in the mini pig. Clin Implant Dent Relat Res. 2012 Aug;14(4):538-45. doi: 10.1111/j.1708-8208.2010.00289.x. Epub 2010 Jun 25. PMID 20586785
- [Background] Kobayashi E, Matsumoto S, Doi H, Yoneyama T, Hamanaka H. Mechanical properties of the binary titanium-zirconium alloys and their potential for biomedical materials. J Biomed Mater Res. 1995 Aug;29(8):943-50. doi: 10.1002/jbm.820290805. PMID 7593037
- [Background] Al-Nawas B, Bragger U, Meijer HJ, Naert I, Persson R, Perucchi A, Quirynen M, Raghoebar GM, Reichert TE, Romeo E, Santing HJ, Schimmel M, Storelli S, ten Bruggenkate C, Vandekerckhove B, Wagner W, Wismeijer D, Muller F. A double-blind randomized controlled trial (RCT) of Titanium-13Zirconium versus Titanium Grade IV small-diameter bone level implants in edentulous mandibles--results from a 1-year observation period. Clin Implant Dent Relat Res. 2012 Dec;14(6):896-904. doi: 10.1111/j.1708-8208.2010.00324.x. Epub 2011 Mar 17. PMID 21414131
- [Background] Benic GI, Gallucci GO, Mokti M, Hammerle CH, Weber HP, Jung RE. Titanium-zirconium narrow-diameter versus titanium regular-diameter implants for anterior and premolar single crowns: 1-year results of a randomized controlled clinical study. J Clin Periodontol. 2013 Nov;40(11):1052-61. doi: 10.1111/jcpe.12156. Epub 2013 Sep 8. PMID 24015975
- [Background] Al-Nawas B, Domagala P, Fragola G, Freiberger P, Ortiz-Vigon A, Rousseau P, Tondela J. A Prospective Noninterventional Study to Evaluate Survival and Success of Reduced Diameter Implants Made From Titanium-Zirconium Alloy. J Oral Implantol. 2015 Aug;41(4):e118-25. doi: 10.1563/AAID-JOI-D-13-00149. Epub 2014 Mar 25. PMID 24666383
- [Background] Quirynen M, Al-Nawas B, Meijer HJ, Razavi A, Reichert TE, Schimmel M, Storelli S, Romeo E; Roxolid Study Group. Small-diameter titanium Grade IV and titanium-zirconium implants in edentulous mandibles: three-year results from a double-blind, randomized controlled trial. Clin Oral Implants Res. 2015 Jul;26(7):831-40. doi: 10.1111/clr.12367. Epub 2014 Apr 9. PMID 24713048
- [Background] Klein MO, Schiegnitz E, Al-Nawas B. Systematic review on success of narrow-diameter dental implants. Int J Oral Maxillofac Implants. 2014;29 Suppl:43-54. doi: 10.11607/jomi.2014suppl.g1.3. PMID 24660189
- [Background] Hammerle CH, Chen ST, Wilson TG Jr. Consensus statements and recommended clinical procedures regarding the placement of implants in extraction sockets. Int J Oral Maxillofac Implants. 2004;19 Suppl:26-8. No abstract available. PMID 15635943
- [Background] Mombelli A, van Oosten MA, Schurch E Jr, Land NP. The microbiota associated with successful or failing osseointegrated titanium implants. Oral Microbiol Immunol. 1987 Dec;2(4):145-51. doi: 10.1111/j.1399-302x.1987.tb00298.x. No abstract available. PMID 3507627
- [Background] Buser D, Martin W, Belser UC. Optimizing esthetics for implant restorations in the anterior maxilla: anatomic and surgical considerations. Int J Oral Maxillofac Implants. 2004;19 Suppl:43-61. PMID 15635945
- [Background] Furhauser R, Florescu D, Benesch T, Haas R, Mailath G, Watzek G. Evaluation of soft tissue around single-tooth implant crowns: the pink esthetic score. Clin Oral Implants Res. 2005 Dec;16(6):639-44. doi: 10.1111/j.1600-0501.2005.01193.x. PMID 16307569
- [Background] Laurell L, Lundgren D. Marginal bone level changes at dental implants after 5 years in function: a meta-analysis. Clin Implant Dent Relat Res. 2011 Mar;13(1):19-28. doi: 10.1111/j.1708-8208.2009.00182.x. PMID 19681932
- [Derived] Walter C, Sagheb K, Blatt S, Klein MO, Herrmann J, Kleinheinz J, Al-Nawas B. Evaluation of the clinical safety and performance of a narrow diameter (2.9 mm) bone-level implant: a 1-year prospective single-arm multicenter study. Int J Implant Dent. 2023 Sep 19;9(1):32. doi: 10.1186/s40729-023-00495-x. PMID 37725234

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First site was initiated on 11th DEC 2015 (Mainz University). The first patient was included on 12 FEB 2016 and the last patient out was on 07 JUN 2019 (last 1-year follow-up). The last centre was closed on 10 DEC 2019 (Münster).
Pre-assignment Details: This was a non-randomized study (N/A).
Period: Overall Study
Arm/Group | BLT Implant Ø 2.9 mm
Started | 46 (First study centre initiation.)
Included | 41
Completed | 38 (Last study centre close-out.)
Not Completed | 8
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 2
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Arm/Group | BLT Implant Ø 2.9 mm
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.53 (18.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 41
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Germany | 41

OUTCOME MEASURES:

1. Primary Outcome: Implant Survival Rate at 12 Months After Implant Placement
Description: A "surviving implant" is an implant stably inserted in the subject's jaw bone at the time of assessment.
Time Frame: 12 months after implant placement
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BLT Implant Ø 2.9 mm
Number analyzed (Participants) | 41
percentage of participants | 92.68 [79.00 to 97.58]

2. Secondary Outcome: Pink Esthetic Score (PES) at 6 Months After Implant Placement
Description: The Pink esthetic score allows an objective evaluation of peri-implant soft tissue of single tooth implants based on 7 variables and is highly reproducible. Each variable will be assessed using a 0-1-2 scoring system; 0 being the lowest, and 2 being the highest value. The minimum achievable PES is 0 and the maximum score is 14. The higher the value, the better the outcome.
Time Frame: 6 months after implant placement
Population: 11 missing values.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | BLT Implant Ø 2.9 mm
Number analyzed (Participants) | 30
score on a scale | 11.2 [10.5 to 11.9]

3. Other Pre Specified Outcome: Implant Success Rate at 12 Months After Implant Placement
Description: A "successful implant" is an implant where all of the following success criteria (according to Buser et al., 1992) apply:
  1. Absence of persisting subjective discomfort such as pain, foreign body perception and/or dysesthesia (painful sensation);
  2. Absence of recurrent peri-implant infection with suppuration;
  3. Absence of tactile implant mobility;
  4. Absence of a continuous peri-implant radiolucency.
Time Frame: 12 months after implant placement
Population: 2 missing values.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BLT Implant Ø 2.9 mm
Number analyzed (Participants) | 39
percentage of participants | 89.7 [75.8 to 97.1]

4. Other Pre Specified Outcome: Marginal Bone Level Changes at 12 Months After Implant Placement
Description: An independent expert is contracted to perform the bone level measurements from the X-rays. The vertical bone level is evaluated by measuring the distance from the implant shoulder to the first visible bone contact on the implant. Measurements are taken at the mesial and distal aspects of the implant, and an average value is calculated. Mean bone level changes are computed by subtracting the average bone level at 12 months after implant placement from the average bone level at baseline (implant placement). Hence, negative bone level changes are representing bone loss; vice versa positive changes representing bone gain. Measurements take into account distortion based on changes on the radiograph from the true dimension of the implant.
Time Frame: Baseline and 12 months after implant placement
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | BLT Implant Ø 2.9 mm
Number analyzed (Participants) | 34
mm | -0.3 [-0.4 to -0.1]

5. Other Pre Specified Outcome: Incidence of Adverse Events and Adverse Device Effects
Description: At each visit the Investigator should determine if any adverse events occurred since the last study visit by speaking with the patient and reviewing any dental and medical records. These AEs, along with any AEs from the current study visit, should be documented and reported as described in Section 8 of the protocol. In addition the Investigator should evaluate the status of any ongoing AEs throughout the study.
Time Frame: Screening, Baseline, 7-14 days after implant placement, 6 weeks after implant placement, 4 months after implant placement, 6 months after implant placement and 12 months after implant placement
Measure: Count of Participants; unit: Participants
Arm/Group | BLT Implant Ø 2.9 mm
Number analyzed (Participants) | 41
Participants
  Adverse Events (AE) | 10
  Adverse Device Effects (ADE) | 6
  Serious Adverse Events | 0
  Serious Adverse Device Effects | 0
  Unanticipated Serious Adv. Device Effect (USADE) | 0
  No AEs | 25

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse Events were recorded at every patient visit and monitored during IMV. Safety Board meetings were conducted to assess the reported and monitored AEs from a Sponsor-Perspective.
Arm/Group | BLT Implant Ø 2.9 mm
All-Cause Mortality (participants affected / at risk) | 0/41
Serious Adverse Events (participants affected / at risk) | 0/41
Other Adverse Events (participants affected / at risk) | 10/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BLT Implant Ø 2.9 mm (N=41)
Implant lost (Surgical and medical procedures) | 3 (3) — Implant lost on pos. 22, subject discontinued.
Common cold (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Inflammation (General disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-09): https://cdn.clinicaltrials.gov/large-docs/66/NCT02699866/Prot_SAP_000.pdf